CLINICAL TRIAL: NCT07154329
Title: Examining the Effect of Internet-Based EMDR Flash Intervention (SKY-Flash) on University Students' Test Anxiety Levels and User Experiences
Brief Title: Internet-Based EMDR Flash Intervention for Test Anxiety in University Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Burak Köksal, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01.10.2024; 16.19
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Test Anxiety
Keywords: Internet-based intervention; EMDR Flash; Psychological Well-Being; University Students; Randomized Controlled Trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, parallel assignment design. University students will be randomly allocated to either the intervention group or the wait-list control group. The intervention group will complete a six-module internet-based EMDR Flash program (SKY-Flash). The control group will not receive any intervention during the study period but will gain access to the program after follow-up assessments. Data will be collected at pre-test, post-test, and one-month follow-up to evaluate the effectiveness and usability of the intervention.
Who Masked: Participant
Masking Description: Participants are blinded to group assignment. They are not informed whether they are in the intervention group or in the wait-list control group. Investigators are aware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Internet-Based EMDR-Flash Program (Experimental): Participants in this group will receive the internet-based EMDR-Flash intervention designed to reduce test anxiety. The program includes structured online sessions where participants apply EMDR-Flash techniques in a unguided digital format.
  Interventions: Behavioral: Internet-Based EMDR-Flash Program
- Wait-list Control Group (No Intervention): Participants assigned to this group will not receive the intervention during the study period. They will remain on a wait-list and will be offered access to the internet-based EMDR-Flash program after the completion of the study.

INTERVENTIONS:
Behavioral: Internet-Based EMDR-Flash Program — Self-guided, internet-based EMDR-Flash program (SKY-Flash) tailored to reduce test anxiety in university students. Delivered via a secure web platform with no live therapist involvement. The intervention comprises six ~40-minute modules completed independently during the study. Each module includes brief psychoeducation and step-by-step EMDR-Flash procedures (focus on a positive engaging image with brief "flash" cues), guided practice, and in-platform exercises. Gamification (progress tracking, badges) and automated prompts support adherence. Unlike CBT-based online programs or clinician-delivered EMDR, this is a fully automated, low-intensity Flash protocol adapted to exam-related distress. Safety messaging and referral resources are embedded; access is via individual login and usage is recorded for adherence.
  Arms: Intervention Group - Internet-Based EMDR-Flash Program

SUMMARY:
The aim of this study is to investigate whether an Internet-based EMDR Flash intervention can help reduce exam anxiety among university students. Participants will utilize the online SKY-Flash program and report their levels of exam anxiety at pre-intervention, post-intervention, and follow-up assessments. In addition, the study will collect feedback regarding participants' overall experiences with the program. The primary objective is to determine whether SKY-Flash constitutes a practical and effective approach to reducing exam anxiety among students, while also exploring their perceptions of the intervention.

DETAILED DESCRIPTION:
Test anxiety is a common problem among university students, often linked to academic pressure, limited access to professional support, and stigma around seeking help. Students with high levels of test anxiety may experience stress, concentration problems, and reduced academic performance. While face-to-face psychological interventions can be effective, many students cannot benefit from them due to financial, logistical, or accessibility barriers.

This study introduces SKY-Flash, an internet-based version of the EMDR Flash technique. The program was designed as a self-help intervention that students can use independently, without therapist guidance. The aim is to reduce test anxiety and improve psychological well-being by adapting EMDR Flash procedures into an online format that is accessible, private, and user-friendly.

The research will be conducted as a randomized controlled trial with two groups: an intervention group and a wait-list control group. A total of 168 university students will be recruited and randomly assigned to one of the groups. Participants in the intervention group will complete a six-module online program based on EMDR Flash principles. The modules include interactive exercises, multimedia elements, and gamification features to support engagement and reduce dropout. The control group will not receive any intervention during the study period but will gain access to the program after follow-up assessments.

Data will be collected at three time points: pre-test, post-test, and one-month follow-up. Primary outcomes will be test anxiety, measured by the Westside Test Anxiety Scale. Secondary outcomes will include psychological well-being and usability feedback. In addition, semi-structured interviews will be conducted with a subgroup of participants to gather in-depth information about usability and user experience.

The study is expected to show whether an online EMDR Flash intervention can effectively reduce test anxiety and improve well-being in university students. If effective, SKY-Flash may serve as a scalable, cost-effective, and stigma-free resource for students who struggle with test anxiety and have limited access to psychological services.

ELIGIBILITY:
Inclusion Criteria:

Voluntary participation in the study Being older than 18 years and currently enrolled as a university student Having a valid e-mail address Having internet access (computer or mobile device) Scoring above the average on the Test Anxiety Scale Scoring below 15 on the Patient Health Questionnaire-9 (PHQ-9), based on established cutoff points

Exclusion Criteria:

Currently receiving psychological help from a psychologist, counselor, or psychiatrist Having any diagnosed psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Test Anxiety (Westside Test Anxiety Scale Scores) | participants will be assessed at baseline (Week 0), immediately after the intervention (Week 6), and again at a follow-up point 10 weeks later
  The primary outcome is the change in test anxiety levels, assessed with the Westside Test Anxiety Scale (WTAS). The WTAS is a validated self-report measure specifically developed to assess test-related anxiety and performance-impairing worry. Higher scores indicating greater test anxiety. This outcome will determine whether the internet-based EMDR-Flash intervention reduces participants' test anxiety compared to the control condition.
Change in Test Anxiety | participants will be assessed at baseline (Week 0), immediately after the intervention (Week 6), and again at a follow-up point 10 weeks later
  The primary outcome is the change in test anxiety levels, assessed with the Westside Test Anxiety Scale (WTAS). The WTAS is a validated self-report measure specifically developed to assess test-related anxiety and performance-impairing worry. . This outcome will determine whether the internet-based EMDR-Flash intervention reduces participants' test anxiety compared to the control condition.

SECONDARY OUTCOMES:
Change in Psychological Well-Being (Psychological Well-Being Scale) | From baseline (Week 0) to post-intervention (Week 6), with follow-up assessments at Week 10.
  Psychological well-being will be measured using the Ryff Psychological Well-Being Scale. The total score reflects overall well-being, with higher scores indicating greater psychological well-being. This outcome will evaluate whether the intervention improves students' well-being in addition to reducing test anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Köksal, Dr., Principal Investigator — Tokat Gaziosmanpaşa University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including demographic information (age, gender, academic year), baseline and follow-up scores on the Test Anxiety Scale, PHQ-9, and WETSIDE measures. No personally identifiable information will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified IPD will be available beginning 6 months after publication of the main results and will be accessible for a period of 5 years
Access Criteria: Data will be made available to qualified researchers affiliated with academic institutions upon reasonable request. Requests will be reviewed by the study team, and data will be shared through secure data transfer agreements ensuring participant confidentiality